CLINICAL TRIAL: NCT03941457
Title: Clinical Research of ROBO1 Specific BiCAR-NK Cells on Patients With Pancreatic Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asclepius Technology Company Group (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AsclepiusTCG03
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-tumor response of BiCAR-NK cells (ROBO1 CAR-NK cells) (Experimental): Patients with relapsed and refractory pancreatic cancer of ROBO1 expression will be treated with BiCAR-NK cells (ROBO1 CAR-NK cells).
  Interventions: Biological: BiCAR-NK cells (ROBO1 CAR-NK cells)

INTERVENTIONS:
Biological: BiCAR-NK cells (ROBO1 CAR-NK cells) — The subject will be observed for any side effects during this time and all the adverse events will be recorded.

SUMMARY:
Immunotherapy has become the major breakthrough and the most promising treatment, with the host of development of tumor biology, molecular biology and immunology. ROBO1 is a potential target and spectacular paradigm in the treatment of solid tumors. This study is for evaluation of the safety and efficacy of ROBO1 CAR-NK cell immunotherapy for pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic pancreatic adenocarcinoma
2. Patients aged between 18 and 75
3. ROBO1 expression in malignancy tissues detected by immuno-histochemistry (IHC)
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Life expectancy greater than 3 months
6. Subjects must have measurable disease as defined by RECIST 1.1 criteria
7. Satisfactory organ and bone marrow function: White blood cell count (WBC) ≥ 3.0×10^9/L, Platelets ≥ 70×10^9/L, Hb ≥ 9.0g/dL, lymphocyte (LY) ≥ 0.7×10^9/L, LY% ≥ 15%, Alb ≥ 2.8g/dL, serum lipase and amylase < 1.5 × upper limit of normal, serum creatinine ≤ 2.5mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5×upper limit of normal, serum total bilirubin ≤ 2.0mg/dL. These tests must be conducted within 7 days prior to registration
8. Karnofsky score ≥ 60
9. Ability to give informed consent

Exclusion Criteria:

1. Previously treated with any gene therapy products
2. Patients who are receiving any other investigational agents
3. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant
4. Active systemic infections (e.g.: requiring anti-infective treatment), coagulation disorders or any other major medical illnesses
5. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease)
6. Concurrent opportunistic infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment related adverse events as assessed by CTCAE v4.03 | 1 year
  Defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, Shanghai Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No